CLINICAL TRIAL: NCT02028845
Title: Loop-tipped Guidewire in Selective Biliary Cannulation: a Prospective, Randomized, Controlled Trial
Brief Title: Loop-tipped Guidewire in Selective Biliary Cannulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Yoo Byung Moo, Assistant Professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AJIRB-DEV-DE2-13-175
Record Dates: First submitted 2013-12-31; First posted 2014-01-07 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Choledocholithiasis; Bile Duct Cancer; Pancreatic Cancer; Ampullary Tumor
MeSH Terms: conditions — Choledocholithiasis; Bile Duct Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Loop guidewire (Active Comparator): This study has two arms. We will compare the performance of a loop-tipped guidewire with a straight-tipped guidewire in achieving successful deep biliary cannulation with loop guidewire.
  Interventions: Device: Biliary cannulation with loop guidewire
- Straight guidewire (Active Comparator): This study has two arms. We will compare the performance of a loop-tipped guidewire with a straight-tipped guidewire in achieving successful deep biliary cannulation with straight guidewire.
  Interventions: Device: Biliary cannulation with straight guidewire

INTERVENTIONS:
Device: Biliary cannulation with loop guidewire — Selective biliary cannulation during endoscopic retrograde cholangiopancreatography
  Arms: Loop guidewire
Device: Biliary cannulation with straight guidewire — Selective biliary cannulation during endoscopic retrograde cholangiopancreatography
  Arms: Straight guidewire

SUMMARY:
1. Background

   * Advanced guidewires with a U-shaped tip could effectively cross the long or multi-occlusive segment smoothly and go into the distal outflow vessel.
   * The guidewire looping technique is a safe and effective method for the recanalization of the occluded lesions in infrapopliteal vessels.
2. Objective - To compare the performance a loop-tipped guidewire with a straight-tipped guidewire in achieving successful deep biliary cannulation.
3. Design

   - Prospective randomized trial.
4. Setting:

   - Tertiary-care medical center
5. Patients

   - This study will involve 192 patients with biliary diseases which require endoscopic retrograde cholangiopancreatography.
6. Intervention - Cannulation of bile duct by using a loop-tipped guidewire or a straight-tipped guidewire
7. Main outcome measurements - Compare the cannulation success rate, the duration of the cannulation, immediate and late complications.

ELIGIBILITY:
Inclusion Criteria:

* age > 19 and ability to consent
* no evidence of significant cardiopulmonary or medical comorbidities precluding participation

Exclusion Criteria:

* Known gastroduodenal anatomic abnormalities
* Coagulation disorders (international normalized ratio > 1.5 or platelet count < 50000 cells/cubic millimeter)
* Prior gastric surgery,endoscopic retrograde cholangiopancreatography
* Pregnancy

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2014-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
The cannulation success rate | Up to 9 months, The primary outcome measure will be assessed after the enrollment of patients (anticipated time: 2014/08/30).

SECONDARY OUTCOMES:
The duration of the cannulation, immediate and late complications. | Up to 9 months, The secondary outcome measure will be assessed after the enrollment of patients (anticipated time: 2014/08/30).

CONTACTS AND LOCATIONS:
Overall Officials: Byung Moo Yoo, MD, PhD, Principal Investigator — Department of Gastroenterology, Ajou University School of Medicine
Locations (1):
- Department of Gastroenterology, Ajou University School of Medicine, Suwon, Gyeonggi-do, South Korea